CLINICAL TRIAL: NCT00885703
Title: A Phase I/II Dose-Finding Study of High-Dose Fluconazole Treatment in AIDS-Associated Cryptococcal Meningitis
Brief Title: High-Dose Fluconazole for the Treatment of Cryptococcal Meningitis in HIV-Infected Individuals
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5225 (HiFLAC); 10149 (Registry Identifier: DAIDS-ES); ACTG A5225; HiFLAC; A5225/HiFLAC; A5225
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2018-02

CONDITIONS: Cryptococcal Meningitis; HIV Infections
Keywords: CM; HIV; Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; Meningitis | interventions — Fluconazole; Amphotericin B; amphotericin B, deoxycholate drug combination; liposomal amphotericin B

STUDY DESIGN:
Intervention Model Description: Phase 1 was the dose escalation phase which used a sequential model. Phase 2 was the dose validation phase which used a parallel model. Analyses combine arms from Phase 1 and Phase 2, as appropriate, for validation.

ARMS (7):
- Stage 1, Fluconazole 1200mg (Experimental): Participants receive Fluconazole 1200mg induction dose in Stage 1
  Interventions: Drug: Fluconazole
- Stage 1, Fluconazole 1600mg (Experimental): Participants receive Fluconazole 1600mg induction dose in Stage 1
  Interventions: Drug: Fluconazole
- Stage 1, Fluconazole 2000mg (Experimental): Participants receive Fluconazole 2000mg induction dose in Stage 1
  Interventions: Drug: Fluconazole
- Stage 1, Ampho B (Active Comparator): Participants receive Amphotericin B followed by Fluconazole in Stage 1
  Interventions: Drug: Fluconazole; Drug: Amphotericin B
- Stage 2, Fluconazole 1600mg (Experimental): Participants receive Fluconazole 1600mg induction dose in Stage 2
  Interventions: Drug: Fluconazole
- Stage 2, Fluconazole 2000mg (Experimental): Participants receive Fluconazole 2000mg induction dose in Stage 2
  Interventions: Drug: Fluconazole
- Stage 2, Ampho B (Active Comparator): Participants receive Amphotericin B followed by Fluconazole in Stage 2
  Interventions: Drug: Fluconazole; Drug: Amphotericin B

INTERVENTIONS:
Drug: Fluconazole — Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
  Other Names: Diflucan
Drug: Amphotericin B — Step 1: [For participants randomized to Ampho B] Ampho B given intravenously for approximately 2 weeks at a dosage of 0.7 to 1.0 mg/kg, dependent on a participant's weight
  Other Names: Amphotericin B deoxycholate; Ampho B; Amphocin; Fungizone; AmBisome; Abelecet; Amphotec
  Arms: Stage 1, Ampho B; Stage 2, Ampho B

SUMMARY:
Cryptococcal meningitis (CM) is an infection of the membranes covering the brain and spinal cord, caused by the fungus Cryptococcus neoformans. CM most often affects people with compromised immune systems, like those with advanced HIV infection. This study explored the safety, tolerability, and therapeutic effect of a new treatment regimen with high-dose fluconazole for management of CM in HIV-infected patients.

DETAILED DESCRIPTION:
CM is the most common central nervous system (CNS) complication of AIDS worldwide and accounts for up to a third of all deaths from AIDS in many developing countries. Current treatments for CM are lacking in both effectiveness and accessibility, particularly in limited-resources settings. Conventional therapies utilizing an amphotericin B deoxycholate (ampho B)-based regimen require maintaining intravenous access (IV) and monitoring and treating any associated complications. The price to acquire ampho B can also be prohibitive to successful treatment. Cumulatively, a treatment course with ampho B is neither cost effective nor administratively efficient, leaving patients either untreated or inadequately treated with low-dose regimens of fluconazole alone.

Fluconazole is widely available, inexpensive, can be given orally, has a demonstrated safety profile over a broad range of doses, and has proven activity against the fungus that causes CM, Cryptococcus neoformans. All of these factors make fluconazole a potential treatment option for a wide range of people. However, at its present recommended dosage, fluconazole is only expected to be successful in 34% to 42% of patients. This rate is lower than regimens combining fluconazole with other treatments including flucytosine or ampho B.

The purpose of this study was to evaluate whether high-dose fluconazole is safe and effective for the treatment of CM for up to 10 weeks. This study also collected information about treating CM with ampho B (either alone or with another drug, either flucytosine or fluconazole).

For this study, 168 HIV-infected people with CM participated for a duration of 24 weeks. This study proceeded with 2 stages and each stage consisted of up to 4 steps. Participants could take part in only one stage of the study. Stage 1 measured the maximum tolerated dose (MTD) of fluconazole in participants. Stage 2 consisted of dose validation and safety monitoring.

In Stage 1, participants were randomly assigned to receive either fluconazole only or an ampho B-based regimen (a regimen that is either ampho B alone or ampho B in combination with 5-fluorocytosine or fluconazole, according to the local standard of care).Three doses of fluconazole were tested, and the MTD was found to be 2000 mg/day. The two higher doses of fluconazole tested in Stage 1 (1600 mg/day and 2000 mg/day doses) were tested further in Stage 2 of the study.

Participants enrolled in Stage 2 were randomly assigned to receive treatment with either fluconazole only (at one of the 2 doses (1600 mg/day or 2000 mg/day) found to be safe in Stage 1) or an ampho B-based regimen.

After randomization in Step 1, participants in both Stage 1 and Stage 2 could be enrolled in up to three additional steps. In Step 2, participants who were randomly assigned to receive the ampho B-based regimen and who were intolerant to the regimen (experienced a treatment limiting toxicity [TLT]) received fluconazole (400-800mg daily). Participants who received study-provided fluconazole in Step 1 or in Step 2 could be enrolled in Step 3 if they had a negative cerebrospinal fluid (CSF) culture. Participants in Step 3 received fluconazole (400mg daily) until Week 10. At Week 10, all participants were enrolled in Step 4 and received a daily dose of fluconazole of 200mg until the end of the study (Week 24). Participants in both stages beginning treatment with ampho B received daily ampho B intravenously for up to 2 weeks.

Before entering the study, potential participants attended a screening visit where they had CSF collected via lumbar puncture. HIV testing was also conducted, along with clinical assessments, and a health and medical history questionnaire. Participants had blood collection, an electrocardiogram (ECG), and a pregnancy test (if applicable) at that visit. Once accepted into the study, participants again answered questions about their health and medication history; had a complete physical exam, blood collection, HIV testing, neurological exam, lumbar puncture, and ECG; and may have had a pregnancy test (if applicable).

Study visits occurred during Weeks 1 (at Days 1, 4, and 7), 2, 4, 6, 8, 10, and 24, and extra visits could occur for individualized reasons. Total study duration was 24 weeks. Plasma, urine, serum, and CSF samples were collected from all participants and stored for possible future use.

Note on efficacy population versus safety population: After entering the study, participants had their CM diagnosis confirmed by testing of the CSF collected via lumbar puncture. Confirmation could take up to 2 weeks after study entry. Due to the mortality rate of CM, participants received treatment before CM diagnosis confirmation. Post-entry 12 participants either reported non-confirmatory baseline results making them ineligible. An additional 2 participants were found to be ineligible for the study but died prior to being found ineligible (one had non-confirmatory baseline results, one was on a disallowed medication) All participants (n=168) are included in the safety population. Participants who were ineligible after study entry were excluded from the efficacy population (n=16). The efficacy population had 154 participants. Outcomes will specify if the efficacy population is used instead of the safety population.

ELIGIBILITY:
Inclusion Criteria - Step 1

* CM documented either by a positive CSF cryptococcal culture, a positive CSF India ink preparation, or a positive CSF cryptococcal antigen latex agglutination test within 7 days prior to entry. More information on this criterion can be found in the protocol.
* CSF collection for quantitative cryptococcal culture within 72 hours prior to study entry or planned to be performed at study entry
* HIV-1 infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by or within 10 days after study entry by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, by HIV-1 antigen, or by plasma HIV-1 RNA viral load. More information on this criterion can be found in the protocol.
* Ability to take oral medications. NOTE: Administration of fluconazole tablets via nasogastric tube is permitted.
* For patients with a co-morbid complication of HIV, including opportunistic infections, reasonable certainty that the site investigator will be able to perform CSF sampling and manage expected study drug toxicities. More information on this criterion can be found in the protocol.
* For female participants of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months [i.e., who have had menses within the preceding 24 months, or have not undergone surgical sterilization, for example, a hysterectomy, or bilateral oophorectomy or salpingotomy]) a negative serum or urine pregnancy test result must be obtained within 2 days prior to study entry
* All participants must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
* If participating in sexual activity that could lead to pregnancy, female study participants must agree to the simultaneous use of two forms of contraception (listed in protocol) during sexual activity, and male study participants must agree to use a condom during such sexual activity. This requirement continues while the study participant is on study treatment and for 6 weeks after fluconazole has been discontinued. More information on this criterion can be found in the protocol.
* Study participants who are not of reproductive potential (defined as women who have been post-menopausal for at least 24 consecutive months, women who have undergone surgical sterilization [e.g., hysterectomy, or bilateral oophorectomy or salpingectomy], or men who have documented azoospermia) are eligible without the requirement to use contraceptives. More information on this criterion can be found in the protocol.
* Willingness and ability to adhere to dose schedules and mandatory procedures
* Measured or calculated creatinine clearance of 50 mL/min or more within 3 days prior to study entry. More information on this criterion can be found in the protocol.
* The following laboratory values within 3 days prior to study entry: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase less than or equal to 5 times the upper limit of normal (ULN); total bilirubin less than or equal to 2.5 times ULN; absolute neutrophil count (ANC) equal to or greater than 750/mm^3; platelet count equal to or greater than 50,000/mm^3; hemoglobin equal to or greater than 7.0 g/dL
* Ability and willingness of the participant or legal guardian/representative to give informed consent
* Availability at the site for at least 2 weeks of its standard-of-care ampho B-based regimen

Exclusion Criteria - Step 1

* Expected survival of 2 weeks or less, in the opinion of the site investigator and, if available, the primary care provider
* For patients with a comorbid complication of HIV, anticipated difficulty, in the opinion of the site investigator, in judging response to study treatment as a result of the comorbid complication or the drugs used to treat it
* Breastfeeding
* A prior episode of CM, either as indicated by patient or as noted in patient medical records
* Use of certain drugs within specified time periods. More information on this criterion can be found in the study protocol.
* For candidates who are currently taking nevirapine, the inability to discontinue nevirapine and replace it with a drug that does not have fluconazole drug interactions at or by study entry in the event they are randomized to a high-dose fluconazole treatment arm. More information on this criterion can be found in the study protocol.
* Known allergy, sensitivity to, or intolerance of fluconazole or other imidazole or triazole compounds or to ampho B or other components of the standard of care ampho B based regimen
* History of clinically significant cardiac disease, in the opinion of the site investigator, including symptoms of ischemia, coronary artery disease, congestive heart failure, or arrhythmia
* ECG with QTc interval greater than 450 msec within 7 days prior to study entry. More information on this criterion can be found in the study protocol.
* History of CNS disorder (excluding mood disorders) or concurrent CNS disorder(s) that, in the opinion of the investigator, would interfere with assessment of efficacy (e.g., ability to perform CSF sampling) such as lymphoma, neurocysticercosis, or toxoplasmosis
* Receipt of investigational drug therapy within 30 days prior to study entry without prior approval of the A5225/HiFLAC core team
* Active drug or alcohol use, dependence, or other conditions that in the opinion of the site investigator would jeopardize the safety of a participant in the study or would render the person unable to comply with the study plan

Inclusion Criteria - Step 2

* Randomization to an ampho B-based regimen in Step 1
* Receipt of at least one dose of ampho B-based regimen in Step 1
* Premature discontinuation of ampho B in response to the occurrence of any treatment-limiting toxicity, as described in Section 5 of the A5225/HiFLAC manual of operations (MOPS)

Exclusion Criteria - Step 2

* Receipt of fluconazole monotherapy in Step 1
* Receipt of 8.4 mg/kg or more of ampho B
* At or beyond Day 17 in Step 1

Inclusion Criteria - Step 3

* For participants in Step 1 who are currently receiving study-provided fluconazole and have no plans to discontinue study treatment (except as noted below), a negative CSF culture after 2 weeks incubation from a sample obtained at or before Week 6 (Days 35-49)
* For participants in Step 1 who are currently receiving an ampho B-based regimen or alternative treatment, completion of approximately 2 weeks of treatment. More information on this criterion can be found in the study protocol.
* For participants in Step 2 who are currently receiving study-provided fluconazole and have no plans to discontinue study treatment, negative CSF culture after 2 weeks incubation from a sample obtained at or before Week 6 (Days 35-49).

Exclusion Criteria - Step 3

* On study treatment beyond Week 10 (Day 77) in Step 1 or Step 2
* Currently off study treatment

Inclusion Criteria - Step 4

- On study treatment at Week 10 (Days 63-77) with no plans to discontinue study treatment

Exclusion Criteria - Step 4

- Currently off study treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-04-16 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umesh G. Lalloo, MD, FRCP, Study Chair — Nelson R. Mandela School of Medicine; Robert A. Larsen, MD, Study Chair — USC School of Medicine
Locations (10):
- University of Southern California CRS, Los Angeles, California, United States
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- Kenya (2):
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Rift Valley
  - Moi University Clinical Research Center (MUCRC) CRS, Eldoret
- San Miguel CRS, Lima, Peru
- South Africa (2):
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
- Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai, Thailand
- Joint Clinical Research Centre (JCRC)/Kampala Clinical Research Site, Kampala, Uganda
- Parirenyatwa CRS, Harare, Zimbabwe

REFERENCES:
- [Background] Bicanic T, Meintjes G, Rebe K, Williams A, Loyse A, Wood R, Hayes M, Jaffar S, Harrison T. Immune reconstitution inflammatory syndrome in HIV-associated cryptococcal meningitis: a prospective study. J Acquir Immune Defic Syndr. 2009 Jun 1;51(2):130-4. doi: 10.1097/QAI.0b013e3181a56f2e. PMID 19365271
- [Background] Pappalardo MC, Szeszs MW, Martins MA, Baceti LB, Bonfietti LX, Purisco SU, Baez AA, Melhem MS. Susceptibility of clinical isolates of Cryptococcus neoformans to amphotericin B using time-kill methodology. Diagn Microbiol Infect Dis. 2009 Jun;64(2):146-51. doi: 10.1016/j.diagmicrobio.2009.02.007. Epub 2009 Apr 2. PMID 19345042
- [Background] Seddon J, Mangeya N, Miller RF, Corbett EL, Ferrand RA. Recurrence of cryptococcal meningitis in HIV-infected patients following immune reconstitution. Int J STD AIDS. 2009 Apr;20(4):274-5. doi: 10.1258/ijsa.2008.008312. PMID 19304977
- [Derived] Lalloo UG, Komarow L, Aberg JA, Clifford DB, Hogg E, McKhann A, Bukuru A, Lagat D, Pillay S, Mave V, Supparatpinyo K, Samaneka W, Langat D, Ticona E, Badal-Faesen S, Larsen RA; ACTG A5225 Team. Higher Dose Oral Fluconazole for the Treatment of AIDS-related Cryptococcal Meningitis (HIFLAC)-report of A5225, a multicentre, phase I/II, two-stage, dose-finding, safety, tolerability and efficacy randomised, amphotericin B-controlled trial of the AIDS Clinical Trials Group. PLoS One. 2023 Feb 13;18(2):e0281580. doi: 10.1371/journal.pone.0281580. eCollection 2023. PMID 36780493
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf?sfvrsn=6
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=10

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on February 19, 2010. The first participant enrolled on April 16, 2010. Stage 1 closed on September 5, 2013. A5225 Stage 2 opened on September 15, 2014 and the first participant enrolled on February 2, 2015. Stage 2 closed on August 19, 2016. Ten sites enrolled participants (1 domestic, 9 international).
Groups:
- Stage 1, Fluconazole 1200mg: Participants receive Fluconazole 1200mg induction dose in Stage 1
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1, Fluconazole 1600mg: Participants receive Fluconazole 1600mg induction dose in Stage 1
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1, Fluconazole 2000mg: Participants receive Fluconazole 2000mg induction dose in Stage 1
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1, Ampho B: Participants receive Amphotericin B followed by Fluconazole in Stage 1
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
  Amphotericin B: Step 1: [For participants randomized to Ampho B] Ampho B given intravenously for approximately 2 weeks at a dosage of 0.7 to 1.0 mg/kg, dependent on a participant's weight
- Stage 2, Fluconazole 1600mg: Participants receive Fluconazole 1600mg induction dose in Stage 2
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 2, Fulconazole 2000mg: Participants receive Fluconazole 2000mg induction dose in Stage 2
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 2, Ampho B: Participants receive Amphotericin B followed by Fluconazole in Stage 2
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
  Amphotericin B: Step 1: [For participants randomized to Ampho B] Ampho B given intravenously for approximately 2 weeks at a dosage of 0.7 to 1.0 mg/kg, dependent on a participant's weight
Period: Overall Study
Arm/Group | Stage 1, Fluconazole 1200mg | Stage 1, Fluconazole 1600mg | Stage 1, Fluconazole 2000mg | Stage 1, Ampho B | Stage 2, Fluconazole 1600mg | Stage 2, Fulconazole 2000mg | Stage 2, Ampho B
Started | 22 | 26 | 24 | 24 | 24 | 24 | 24
Completed | 12 | 16 | 13 | 15 | 12 | 11 | 18
Not Completed | 10 | 10 | 11 | 9 | 12 | 13 | 6
Not completed — Death | 9 | 7 | 8 | 7 | 7 | 8 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Ineligible (no CM) | 1 | 3 | 2 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Stage 2, Fluconazole 2000mg: Participants receive Fluconazole 2000mg induction dose in Stage 2
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Total: Total of all reporting groups
Arm/Group | Stage 1, Fluconazole 1200mg | Stage 1, Fluconazole 1600mg | Stage 1, Fluconazole 2000mg | Stage 1, Ampho B | Stage 2, Fluconazole 1600mg | Stage 2, Fluconazole 2000mg | Stage 2, Ampho B | Total
Number analyzed (Participants) | 22 | 26 | 24 | 24 | 24 | 24 | 24 | 168
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.5 [36 to 47] | 33 [28 to 39] | 38 [31 to 48] | 35.5 [30 to 41] | 32.5 [29.5 to 35.5] | 33.5 [29 to 38] | 37.5 [34 to 40] | 36 [30 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 14 | 11 | 10 | 10 | 9 | 78
  Male | 12 | 12 | 10 | 13 | 14 | 14 | 15 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 12 | 21 | 22 | 19 | 24 | 22 | 23 | 143
  Hispanic (regardless of Race) | 0 | 4 | 2 | 1 | 0 | 2 | 1 | 10
  Asian, Pacific Islander | 10 | 1 | 0 | 4 | 0 | 0 | 0 | 15
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 4
  South Africa | 1 | 6 | 3 | 5 | 2 | 3 | 6 | 26
  Uganda | 0 | 2 | 11 | 5 | 14 | 13 | 12 | 57
  Zimbabwe | 2 | 4 | 1 | 3 | 4 | 1 | 3 | 18
  Kenya | 8 | 9 | 7 | 6 | 4 | 6 | 2 | 42
  Thailand | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  Peru | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 6
  India | 5 | 1 | 0 | 3 | 0 | 0 | 0 | 9
Weight [Median (Inter-Quartile Range); unit: kilograms] | 46.5 [42.0 to 52.2] | 50.5 [44.0 to 65.0] | 51.9 [43.5 to 58.5] | 56.8 [47.5 to 64.1] | 49.8 [44.5 to 60.0] | 55.0 [51.6 to 59.1] | 52.5 [48.5 to 60.1] | 52.0 [44.7 to 59.3]
BMI (Body Mass Index) [Median (Inter-Quartile Range); unit: kg/m^2] | 17.2 [15.6 to 19.6] | 19.6 [17.3 to 21.8] | 18.3 [17.2 to 22.7] | 19.8 [16.3 to 24.3] | 18.7 [17.1 to 20.3] | 19.8 [18.6 to 22.5] | 19.6 [17.5 to 22.9] | 18.9 [16.9 to 21.9]
CD4+ [Count of Participants; unit: Participants]
  < 50 cells/mm^3 | 15 | 10 | 17 | 17 | 20 | 16 | 17 | 112
  50 - <100 cells/mm^3 | 6 | 9 | 4 | 4 | 3 | 5 | 5 | 36
  100 - <200 cells/mm^3 | 1 | 4 | 3 | 2 | 0 | 3 | 2 | 15
  200+ cells/mm^3 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 5
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10(copies/mL)] | 5.3 [5.1 to 6.0] | 5.6 [5.1 to 5.8] | 5.5 [5.2 to 5.9] | 5.4 [5.2 to 5.7] | 5.2 [4.9 to 5.5] | 4.9 [2.8 to 5.4] | 4.6 [3.5 to 5.5] | 5.3 [4.7 to 5.7]
Glasgow Coma Score [Count of Participants; unit: Participants] — The Glasgow Coma Score provides an assessment of impairment of conscious level in response to defined stimuli. The GCS is on a scale from 0=worst to 15=best. Population: One participant missing baseline Glasgow Coma Score.
  Participants
    number analyzed (Participants) | 22 | 26 | 24 | 24 | 24 | 23 | 24 | 167
    GCS <15 | 5 | 3 | 5 | 1 | 2 | 0 | 0 | 16
    GCS =15 | 17 | 23 | 19 | 23 | 22 | 23 | 24 | 151
Quantitative Cryptococcal Meningitis Culture [Median (Inter-Quartile Range); unit: Log10 CFU/mL] | 5.18 [4.23 to 6.02] | 4.45 [3.98 to 5.09] | 5.15 [4.25 to 5.80] | 4.37 [3.33 to 5.23] | 5.34 [4.31 to 5.47] | 4.29 [2.05 to 5.32] | 5.14 [3.40 to 5.42] | 5.04 [3.80 to 5.42]
Anti-Retroviral Therapy (ART) Status [Count of Participants; unit: Participants]
  On ART | 0 | 0 | 0 | 0 | 8 | 12 | 11 | 31
  Not on ART | 22 | 26 | 24 | 24 | 16 | 12 | 13 | 137
Opportunistic Infections [Count of Participants; unit: Participants]
  One or more opportunistic infections | 10 | 7 | 11 | 10 | 11 | 9 | 10 | 68
  No opportunistic infections | 12 | 19 | 13 | 14 | 13 | 15 | 14 | 100
Mini Mental Status [Median (Inter-Quartile Range); unit: Scores on a scale] — The Mini Mental Status is a 26-point questionnaire that is used to measure cognitive impairment. Scale is 0=worst to 26=best. Population: Not all participants were able to complete a Mini Mental Status at baseline.
  Scores on a scale
    number analyzed (Participants) | 19 | 25 | 21 | 22 | 23 | 24 | 24 | 158
    (all) | 26 [23 to 26] | 25 [23 to 26] | 26 [22 to 26] | 26 [24 to 26] | 26 [21 to 26] | 26 [19 to 26] | 25.5 [20 to 26] | 26 [22 to 26]
Opening Pressure (from Lumbar Pucture) [Median (Inter-Quartile Range); unit: mm H20] — Population: Not all participants were able to have a lumbar puncture at entry.
  mm H20
    number analyzed (Participants) | 21 | 26 | 23 | 23 | 24 | 24 | 24 | 165
    (all) | 200 [105 to 300] | 200 [150 to 290] | 350 [180 to 550] | 190 [120 to 300] | 200 [150 to 254] | 190 [120 to 235] | 303 [250 to 485] | 210 [141 to 320]
White Blood Cell count (from CSF) [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Not all participants were able to have a lumbar puncture. Of those that did, not all were able to have enough fluid collected for WBC count.
  cells/mm^3
    number analyzed (Participants) | 19 | 21 | 23 | 21 | 23 | 23 | 23 | 153
    (all) | 80 [30 to 500] | 30 [4 to 100] | 17 [9 to 310] | 26 [15 to 133] | 19 [8 to 33] | 16 [12 to 89] | 13 [8 to 53] | 19 [9 to 100]
Albumin [Median (Inter-Quartile Range); unit: g/dL] — Population: Not all participants had an albumin measurement.
  g/dL
    number analyzed (Participants) | 22 | 26 | 24 | 24 | 24 | 23 | 24 | 167
    (all) | 3.0 [2.6 to 3.3] | 3.2 [3.1 to 3.6] | 3.3 [2.9 to 3.6] | 3.2 [2.8 to 3.6] | 3.1 [2.8 to 3.2] | 3.1 [2.7 to 3.6] | 3.1 [2.7 to 3.6] | 3.2 [2.8 to 3.5]
ALT (Alanine Aminotransferase) [Median (Inter-Quartile Range); unit: U/L] | 15.7 [11.0 to 22.8] | 19.0 [13.0 to 29.2] | 24.7 [14.0 to 41.8] | 21.5 [11.7 to 32.7] | 25.2 [17.4 to 38.0] | 24.1 [14.5 to 32.1] | 18.1 [14.5 to 35.3] | 20.6 [14.0 to 32.6]
Creatinine Clearance [Mean (Inter-Quartile Range); unit: mL/min] | 94.2 [79.5 to 112.1] | 94.5 [79.3 to 106.3] | 94.2 [72.7 to 115.2] | 102.3 [81.9 to 135.5] | 94.0 [68.2 to 104.0] | 98.8 [67.3 to 121.8] | 94.4 [77.6 to 113.5] | 95.0 [75.0 to 113.3]
Cryptococcal Antigen (CrAG) Titer [Median (Inter-Quartile Range); unit: titers] — Population: Not all participants had a CrAG titer observed at baseline.
  titers
    number analyzed (Participants) | 22 | 23 | 22 | 23 | 23 | 23 | 22 | 158
    (all) | 756 [256 to 8192] | 128 [32 to 1024] | 815.5 [125 to 8192] | 1050 [160 to 4096] | 256 [20 to 1024] | 128 [16 to 2048] | 416 [128 to 4096] | 452.5 [32 to 2405]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued Study-provided High Dose Fluconazole or Ampho B
Description: Discontinuation of study-provided high dose fluconazole at or by week 10 Discontinuation of study-provided ampho B at or by week 2
  Discontinuation includes discontinuing for any reason, including progression of symptoms, death, etc.
Time Frame: Measured from study entry through Week10
Population: Analysis in safety population (see study detailed description for details)
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Fluconazole 1200mg | Stage 1, Fluconazole 1600mg | Stage 1, Fluconazole 2000mg | Stage 1, Ampho B | Stage 2, Fluconazole 1600mg | Stage 2, Fluconazole 2000mg | Stage 2, Ampho B
Number analyzed (Participants) | 22 | 26 | 24 | 24 | 24 | 24 | 24
Participants | 14 | 11 | 11 | 6 | 12 | 13 | 6
Statistical Analysis 1: Comparison: Stage 1, Fluconazole 1200mg vs Stage 1, Fluconazole 1600mg vs Stage 1, Fluconazole 2000mg vs Stage 1, Ampho B vs Stage 2, Fluconazole 1600mg vs Stage 2, Fluconazole 2000mg vs Stage 2, Ampho B; Testing discontinuation of any dose Fluconazole (pooled by treatment and dose) versus discontinuation of Ampho B (pooled). The null hypothesis is the two treatments have the same proportion of discontinuation; Test type: Superiority; p = 0.0012, Chi-squared — Analysis did not adjust for multiple comparisons

2. Primary Outcome: Categorized Quantitative Culture Results
Description: Count of participants who were CM negative (had no cryptococcal growth), CM negative after switching treatment (switched from Fluconazole to Ampho B or vice versa and later became CM negative), CM positive, Died, Lost to follow-up. Note: CM positive means continued to have cryptococcal growth.
Time Frame: At entry, Week 2, and Week 10
Population: Arms pooled by dose. Analysis in efficacy population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Groups:
- Fluconazole 1200mg: Participants receive Fluconazole 1200mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Fluconazole 1600mg: Participants receive Fluconazole 1600mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Fluconazole 2000mg: Participants receive Fluconazole 2000mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Ampho B: Participants receive Amphotericin B followed by Fluconazole
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
  Amphotericin B: Step 1: [For participants randomized to Ampho B] Ampho B given intravenously for approximately 2 weeks at a dosage of 0.7 to 1.0 mg/kg, dependent on a participant's weight
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 20 | 45 | 43 | 46
Participants
  Week 0: CM Positive | 20 | 45 | 43 | 46
  Week 0: CM Negative | 0 | 0 | 0 | 0
  Week 0: CM Negative after switching treatment | 0 | 0 | 0 | 0
  Week 0: Died | 0 | 0 | 0 | 0
  Week 0: Lost to Follow-up | 0 | 0 | 0 | 0
  Week 2: CM Positive | 12 | 27 | 27 | 29
  Week 2: CM Negative | 3 | 12 | 10 | 13
  Week 2: CM Negative after switching treatment | 0 | 0 | 0 | 0
  Week 2: Died | 5 | 6 | 6 | 4
  Week 2: Lost to Follow-up | 0 | 0 | 0 | 0
  Week 10: CM Positive | 3 | 4 | 3 | 2
  Week 10: CM Negative | 8 | 24 | 22 | 37
  Week 10: CM Negative after switching treatment | 1 | 4 | 5 | 1
  Week 10: Died | 8 | 10 | 12 | 5
  Week 10: Lost to Follow-up | 0 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Fluconazole 1200mg vs Fluconazole 1600mg vs Fluconazole 2000mg vs Ampho B; Among 4 treatment arms, comparison of three categorical groups: (CM negative, CM negative after switching treatment, and CM Positive/Died/Lost to Follow-up) at week 10. The null hypothesis is the 4 treatment arms have no differences at week 10; Test type: Superiority; p = 0.012, Fisher Exact

3. Primary Outcome: Change in Log10 Quantitative CSF Culture Results
Description: Change in quantitative CSF (cerebrospinal fluid) cultures.
  Note: No further CSF specimens are drawn following a negative culture. Thus, only week 2 CSF cultures are considered in this analysis.
Time Frame: Entry and Week 2
Population: Arms pooled by dose. Analysis done in efficacy population (see study detailed description for details). Excludes participants who did not have a week 2 observation.
Measure: Median (Inter-Quartile Range); unit: Log10 CFU/mL
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 15 | 36 | 37 | 40
Log10 CFU/mL | -1.51 [-2.90 to -0.91] | -2.51 [-4.00 to -1.44] | -1.78 [-3.24 to -1.00] | -2.81 [-4.09 to -1.92]
Statistical Analysis 1: Comparison: Fluconazole 1200mg vs Fluconazole 1600mg vs Fluconazole 2000mg vs Ampho B; Comparison of change in quantitative CSF culture among 4 treatment arms. The null hypothesis is the 4 treatment arms have the same change in CSF culture from entry to week 2; Test type: Superiority; p = 0.019, Kruskal-Wallis

4. Primary Outcome: Kaplan Meier (KM) Proportion of Participant Mortality
Description: Kaplan Meier Proportion of participants who died over study with 90% Confidence Intervals.
Time Frame: Measured from study entry through Week 24
Population: Arms pooled by dose in the safety population (see study detailed description for details).
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
proportion of participants | 0.41 [0.26 to 0.60] | 0.30 [0.20 to 0.43] | 0.36 [0.25 to 0.49] | 0.24 [0.15 to 0.36]
Statistical Analysis 1: Comparison: Fluconazole 1200mg vs Ampho B; Comparison of survival from entry to week 24 between Fluconazole 1200mg arm and Ampho B arm. The null hypothesis is there is no difference in survival between these two arms; Test type: Superiority; p = 0.0894, Log Rank — Analysis did not adjust for multiple comparisons
Statistical Analysis 2: Comparison: Fluconazole 1600mg vs Ampho B; Comparison of survival from entry to week 24 between Fluconazole 1600mg arm and Ampho B arm. The null hypothesis is there is no difference in survival between these two arms; Test type: Superiority; p = 0.4828, Log Rank — Analysis did not adjust for multiple comparisons
Statistical Analysis 3: Comparison: Fluconazole 2000mg vs Ampho B; Comparison of survival from entry to week 24 between Fluconazole 2000mg arm and Ampho B arm. The null hypothesis is there is no difference in survival between these two arms; Test type: Superiority; p = 0.1766, Log Rank — Analysis did not adjust for multiple comparisons

5. Secondary Outcome: Results of the Neurological Examination
Description: Results from Glasgow Coma Score, which provides assessment of impairment of conscious level in response to defined stimuli. Min score of 0 and max score of 15 (no mental impairment).
Time Frame: Measured at study entry, Week 2, and Week 10
Population: Arms pooled by dose. Safety population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
Participants
  Week 0: number analyzed (Participants) | 22 | 50 | 47 | 48
  Week 0: Score < 15 | 5 | 5 | 5 | 1
  Week 0: Score = 15 | 17 | 45 | 42 | 47
  Week 2: number analyzed (Participants) | 17 | 42 | 40 | 43
  Week 2: Score < 15 | 2 | 4 | 4 | 5
  Week 2: Score = 15 | 15 | 38 | 36 | 38
  Week 10: number analyzed (Participants) | 12 | 34 | 27 | 34
  Week 10: Score < 15 | 1 | 1 | 1 | 0
  Week 10: Score = 15 | 11 | 33 | 26 | 34

6. Secondary Outcome: Results of Functional Status Evaluation
Description: Functional assessment of work status and ability. Consists of 2 measures: 1) Does participants have full time work status 2) Does participant have functional ability to work.
  The measure from 6 week before enrollment will be referred to as 'baseline'.
Time Frame: Measured 6 weeks before enrollment, at study entry, at Week 10, and at Week 24
Population: Arms pooled by dose. Safety population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
Participants
  Baseline Had full time work status: number analyzed (Participants) | 21 | 50 | 48 | 48
  Baseline Had full time work status | 18 | 41 | 36 | 42
  Entry Had full time work status: number analyzed (Participants) | 21 | 50 | 48 | 48
  Entry Had full time work status | 3 | 9 | 8 | 9
  Week 10 Had full time work status: number analyzed (Participants) | 12 | 32 | 27 | 34
  Week 10 Had full time work status | 3 | 16 | 9 | 13
  Week 24 Had full time work status: number analyzed (Participants) | 12 | 30 | 23 | 33
  Week 24 Had full time work status | 7 | 18 | 17 | 22
  Baseline Had functional ability to work: number analyzed (Participants) | 21 | 50 | 48 | 48
  Baseline Had functional ability to work | 16 | 41 | 32 | 38
  Entry Had functional ability to work: number analyzed (Participants) | 21 | 50 | 48 | 48
  Entry Had functional ability to work | 1 | 8 | 3 | 7
  Week 10 Had functional ability to work: number analyzed (Participants) | 12 | 32 | 27 | 34
  Week 10 Had functional ability to work | 4 | 18 | 9 | 15
  Week 24 Had functional ability to work: number analyzed (Participants) | 12 | 30 | 23 | 33
  Week 24 Had functional ability to work | 7 | 19 | 16 | 24

7. Secondary Outcome: Length of Hospitalization
Description: Duration of first hospitalization in days starting at entry in safety population.
Time Frame: Measured from study entry through Week 10
Population: Arms pooled by dose in safety population (see study detailed description for details). Fluconazole 2000mg arm had one participant data missing (was not admitted to hospital at study entry).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 47 | 48
Days | 15 [10 to 21] | 17.5 [10 to 28] | 18 [13 to 36] | 18.5 [17 to 26]

8. Secondary Outcome: Number of Hospital Admissions
Description: Count of number of times a participant was admitted to the hospital.
Time Frame: Measured from study entry through Week 24
Population: Arms pooled by dose in safety population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
Participants
  1 hospital admission | 18 | 39 | 41 | 37
  2 hospital admissions | 1 | 9 | 6 | 10
  3 hospital admissions | 3 | 2 | 1 | 1

9. Secondary Outcome: Number of Participants With Progression of Symptoms
Description: Progression of symptoms is defined as:
  * Died (including early deaths)
  * Discontinued Fluconazole and started ampho B
  * Had a positive cryptococcal culture at week 10
  * Microbiological Failure (i.e., relapse of CM)
  * Complication of CM (e.g., obstructive hydrocephalus or vascular complications such as venous or arterial thrombosis)
  * CM IRIS causing increased inflammation after ART exposure
  * New CNS Ol (e.g., toxoplasmosis, PML, CNS lymphoma)
  * Possibly related to CM but mechanism indeterminate
  * Other defined complication unrelated to CM
Time Frame: Measured from study entry through Week 24
Population: Arms pooled by dose. Analysis done in efficacy population (see detailed study description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 20 | 45 | 43 | 46
Participants | 14 | 21 | 24 | 19

10. Secondary Outcome: Number of Participants With CNS IRIS
Description: Number of participants who were diagnosed with CNS immune reconstitution inflammatory syndrome (IRIS)
Time Frame: Measured from study entry through Week 24
Population: Arms pooled by dose in study population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
Participants | 1 | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Grade 3 and 4 Adverse Events
Description: Occurrence of grade 3 (severe) and 4 (life-threatening) sign and symptoms events (as defined by FSTRF Appendix 29)
  Occurrence of grade 3 (severe) and 4 (life-threatening) laboratory events (as defined by FSTRF Appendix 76)
  See DAIDS AE Grading table V1.0
Time Frame: Measured from study entry through Week 24
Population: Arms pooled by dose in safety population (see study detailed description for details).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole 1200mg | Fluconazole 1600mg | Fluconazole 2000mg | Ampho B
Number analyzed (Participants) | 22 | 50 | 48 | 48
Participants
  Sign/Symptom Events | 16 | 23 | 32 | 24
  Laboratory Events | 12 | 27 | 26 | 30

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from study entry until end of study (24 weeks).
Description: The protocol required reporting of all Grade >= 3 signs/symptoms, all Grade >= 2 laboratory toxicities, all estimated creatinine clearance values, and all signs/symptoms or laboratory toxicities that lead to a change in treatment, regardless of grade, were recorded. All diagnoses were recorded.
  The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (http://rsc.tech-res.com/safetyandpharmacovigilance/)
Groups:
- Stage 1: 1200mg Fluconazole: Participants receive Fluconazole 1200mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1: 1600mg Fluconazole; Stage 2: 1600mg Fluconazole: Participants receive Fluconazole 1600mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1: 2000mg Fluconazole; Stage 2: 2000mg Fluconazole: Participants receive Fluconazole 2000mg induction dose
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
- Stage 1: Ampho B; Stage 2: Ampho B: Participants receive Amphotericin B followed by Fluconazole
  Fluconazole: Step 1: [For participants randomized to Fluconazole] Induction dose of daily treatment of fluconazole given orally (adjusted according to weight).
  Step 2: [For participants randomized to Ampho B only] If participant is intolerant to Ampho B, participant transitions to fluconazole dosage of 400-800mg daily given orally.
  Step 3: If participant has a negative culture before week 10, participant transitions to consolidation therapy at dosage of 400mg daily given orally.
  Step 4: At week 10, participant transitions to maintenance therapy at dosage of 200mg daily given orally.
  Amphotericin B: Step 1: [For participants randomized to Ampho B] Ampho B given intravenously for approximately 2 weeks at a dosage of 0.7 to 1.0 mg/kg, dependent on a participant's weight
Arm/Group | Stage 1: 1200mg Fluconazole | Stage 1: 1600mg Fluconazole | Stage 1: 2000mg Fluconazole | Stage 1: Ampho B | Stage 2: 1600mg Fluconazole | Stage 2: 2000mg Fluconazole | Stage 2: Ampho B
All-Cause Mortality (participants affected / at risk) | 9/22 | 7/26 | 8/24 | 7/24 | 7/24 | 8/24 | 4/24
Serious Adverse Events (participants affected / at risk) | 14/22 | 13/26 | 13/24 | 11/24 | 10/24 | 12/24 | 6/24
Other Adverse Events (participants affected / at risk) | 22/22 | 26/26 | 24/24 | 24/24 | 24/24 | 24/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: 1200mg Fluconazole (N=22) | Stage 1: 1600mg Fluconazole (N=26) | Stage 1: 2000mg Fluconazole (N=24) | Stage 1: Ampho B (N=24) | Stage 2: 1600mg Fluconazole (N=24) | Stage 2: 2000mg Fluconazole (N=24) | Stage 2: Ampho B (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disseminated cryptococcosis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 5 | 7 | 6 | 2 | 5 | 2 | 4
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: 1200mg Fluconazole (N=22) | Stage 1: 1600mg Fluconazole (N=26) | Stage 1: 2000mg Fluconazole (N=24) | Stage 1: Ampho B (N=24) | Stage 2: 1600mg Fluconazole (N=24) | Stage 2: 2000mg Fluconazole (N=24) | Stage 2: Ampho B (N=24)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 3 | 1 | 3 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 2 | 0
Anorectal swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 4 | 5 | 5 | 6 | 5
Asthenia (General disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0
Chest pain (General disorders) | 3 | 2 | 1 | 2 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 2 | 0 | 1 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 4 | 2 | 10 | 5 | 5
Pyrexia (General disorders) | 7 | 6 | 7 | 8 | 6 | 4 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 2 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 1 | 1
Encephalitis cytomegalovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 3
Malaria (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 6 | 8 | 9 | 10 | 6 | 8 | 5
Meningitis tuberculous (Infections and infestations) | 1 | 1 | 3 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 3 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 2 | 0 | 2 | 0 | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 | 0 | 1 | 1 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 1 | 2 | 2 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 2 | 2 | 2 | 0 | 2 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 4 | 5 | 6 | 3 | 4 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 5 | 9 | 7 | 6 | 3 | 6
Blood albumin decreased (Investigations) | 19 | 18 | 18 | 19 | 19 | 17 | 21
Blood alkaline phosphatase increased (Investigations) | 4 | 2 | 7 | 1 | 5 | 2 | 5
Blood bicarbonate decreased (Investigations) | 4 | 9 | 16 | 6 | 10 | 14 | 10
Blood bilirubin increased (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 2
Blood calcium decreased (Investigations) | 2 | 0 | 1 | 1 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 2 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 5 | 4 | 8 | 12 | 7 | 5 | 13
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1
Blood glucose increased (Investigations) | 12 | 7 | 9 | 7 | 6 | 8 | 8
Blood magnesium decreased (Investigations) | 5 | 0 | 4 | 8 | 2 | 3 | 9
Blood phosphorus decreased (Investigations) | 1 | 0 | 2 | 3 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 14 | 7 | 10 | 13 | 6 | 9 | 13
Blood potassium increased (Investigations) | 2 | 0 | 1 | 2 | 0 | 3 | 2
Blood pressure increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 19 | 21 | 21 | 20 | 18 | 18 | 22
Haemoglobin decreased (Investigations) | 8 | 11 | 9 | 11 | 8 | 8 | 17
Neutrophil count decreased (Investigations) | 4 | 8 | 11 | 6 | 14 | 8 | 10
Platelet count decreased (Investigations) | 7 | 5 | 7 | 5 | 8 | 5 | 5
Weight decreased (Investigations) | 1 | 0 | 2 | 0 | 1 | 4 | 1
White blood cell count decreased (Investigations) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Abnormal loss of weight (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 4 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1 | 2 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 3 | 0 | 2 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 4 | 4 | 8 | 6 | 7 | 5 | 7
Seizure (Nervous system disorders) | 2 | 2 | 2 | 4 | 2 | 3 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 4 | 2 | 4 | 4 | 0 | 3 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 1 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 6 | 3 | 3 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 4 | 1 | 1 | 3 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 1
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.